CLINICAL TRIAL: NCT04825002
Title: Detection of Clinically Significant Prostate Cancer Using a Urinary Multimarker Sensor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Biomaterials Research Center, Korea Institute of Science and Technology (KIST), Seoul, Republic of Korea (Unknown); Korea Medial Device Development Fund grant funded by the Korean government (Unknown)
Responsible Party: Principal Investigator, In Gab Jeong, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0305
Record Dates: First submitted 2021-03-20; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; biopsy; urine; biomarker; nanoparticle
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urinary multimarker sensor arm (Experimental): A urine of this group will be collected and measured using a newly developed urinary multimarker sensor (ANXA3, PSMA, ERG, ENG)
  Interventions: Diagnostic Test: Urinary multimarker sensor

INTERVENTIONS:
Diagnostic Test: Urinary multimarker sensor — We will develop a urinary multimarker sensor, able to measure trace amounts of biomarkers from naturally voided urine.

SUMMARY:
This trial aims to develop and validate the urinary multimarker sensor which can measure trace amounts of biomarkers from naturally voided urine in men referred with clinical suspicion of prostate cancer who have had no prior prostate biopsy. The investigators hypothesize that urinary multimarker sensor will help to avoid unnecessary prostate biopsy while detect the clinically significant cancers.

DETAILED DESCRIPTION:
The investigators will develop a urinary multimarker sensor, able to measure trace amounts of biomarkers from naturally voided urine.

1. Urine specimen collection. This study was approved by the Institutional Review Board of the Asan Medical Center (Seoul, Republic of Korea) and informed consent will be obtained from all subjects. Biomarkers diffused passively from prostate tissue to the urethra and will be collected from naturally voided urine. Urine will be collected in a sterilized specimen cup containing 10 vol% RNA stabilizer and 1vol% antibiotics and stored in a refrigerator for less than a week before shipping the sample to the laboratory
2. To measure the electrical signals from the four different biomarkers in the urine, the four sensing channels in the extended gate of an field-effect transistor biosensor will be conjugated to antibodies, thus capturing different biomarkers.
3. Without any pretreatment, urine will be added directly to the four different sensing channels. After 20 min of reaction time in the four channels, the bottom gate voltage shifts will be measured at the reference current (1 nA). Each urine sample will generate four independent sensing signals from the corresponding biomarkers. The set of sensing signals collected for each patient will be then analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Men undergoing a first-time prostate biopsy to rule out cancer
2. Serum PSA ≥3ng/mL, ≤20ng/mL
3. Age≥50 years, ≤80 years
4. Clinical stage ≤T2c
5. Patients must be able to provide written informed consent.

Exclusion Criteria:

1. Patients has any prior needle biopsy of the prostate
2. Patients has a prior history of prostate cancer
3. Patients has a prior history of pelvic radiation therapy or androgen deprivation therapy
4. Patients has a prior history of BPH operation
5. Patient with uncorrectable coagulopathies
6. Unable to tolerate a TRUS guided biopsy.
7. Patients had 5-alpha reductase inhibitor in the past six months.
8. The patient has had a urinary tract infection or acute prostatitis in the last three months.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-03-22 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence vs. absence of clinically significant prostate cancer on prostate biopsy | through study completion, an average of 3 year
  (≥Gleason score 3+4)

SECONDARY OUTCOMES:
Presence vs. absence of overall prostate cancer | through study completion, an average of 3 year
  presence or absence of prostate cancer at prostate biopsy
Optimal cutoff points for the each biomarker | through study completion, an average of 3 year
  cutoff points for each biomarker (ANXA3, PSMA, ERG, ENG)
Accuracy of each biomarker | through study completion, an average of 3 year
  sensitivity, specificity, positive/negative predictive value
Area Under Curve (Receiver operating curve) by multivariable linear regression model | through study completion, an average of 3 year
  Area Under Curve for each biomarker alone or combination

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No